CLINICAL TRIAL: NCT02913885
Title: Comparative Study Using Biomimetic Remineralization Versus Fluoride Varnish In Management Of White Spot Lesion In Post Orthodontic Treated Patient: (Split Mouth Technique ) A Randomized Clinical Trial
Brief Title: Effect of Curodont Repair on Color Change of White Spot Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aalaa Mohamed Nabil, assistant lecturer, conservative Dentistry Department MTI university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-199
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Active Comparator): curodont repair is a biomimetic regeneration scaffold for remineralization
  Interventions: Drug: Curodont Repair; Drug: fluoride varnish
- Group 1 (Experimental): fluoride varnish inhibit progression of white spot lesion
  Interventions: Drug: Curodont Repair; Drug: fluoride varnish

INTERVENTIONS:
Drug: Curodont Repair — composed of biomimetic regeneration scaffold self-assembling peptides (P11-4) used for remineralization
  Other Names: CURODONT™ REPAIR,Credentis, Switzerland
Drug: fluoride varnish — fluoride inhibit the progression of white spot lesion
  Other Names: 2.26% F, Duraphat, WoelmPharma GmbH, Germany

SUMMARY:
The aim of this study is to compare the effect of color change between remineralizing agent and guided enamel regeneration in treatment of white spot lesion after orthodontic treatments

DETAILED DESCRIPTION:
Roles and responsibilities:

1. Aalaa Mohamed Nabil Amin Abdullatif (A.N.) Operator, data enterer and corresponding author; Assistant lecturer, Conservative Dentistry Department, ModernTechnology University, Egypt.
2. Mohamed Riad (M.R) Main supervisor, data monitoring, auditing Professor, Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
3. Rasha Haridy (R.H.) Co-supervisor, data entry and auditing; Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
4. Ahmed Refaat Mohamed (A.R.) Outcome assessors and data collection; Lecturers, Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
5. Heba fathy (H.F) Outcome assessors and data collection; Assistant lecturer,, Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
6. Ahmed Mamdouh Ahmed (A.M.) Base line data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants' consents; Resident, Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
7. Eman Desouky (E.D.) Sample size calculation; Statistician, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
8. Evidence Based Dentistry Committee (CEBD) Help in reporting study protocol following SPIRIT guidelines; Faculty of Oral and Dental Medicine, Cairo University, Egypt.
9. Research Ethics Committee (CREC) Protocol reviewer of the clinical trial in order to protect the right, safety, dignity and well-being of the participants; Faculty of Oral and Dental Medicine, Cairo University, Egypt.

1-Intervention: A.N. will treat the lesion with 2 % NaOCl for 20 sec, then rinsed and dried. A.N. will etch the lesion with 35 % Phosphoric acid for 20 sec to open up the pores to the subsurface lesion and sub¬sequently rinsed with water for 20 sec and air-dried. A.N. will apply (CURODONT™ REPAIR,Credentis, Switzerland) for two to three minutes. A.N. will advise the patients to rinse the quadrant containing the treated teeth using chlorhexidine mouthwash (Corsodyl, Herrenberg, Germany) until Day 4 and avoid teeth brushing. At D4, A.N. will ask the patients to use a soft tooth brush and tooth paste until Day 8. At this point they will be reverted to their normal oral hygiene procedures.

2-Comparator: A.N. will apply (2.26% F, Duraphat, WoelmPharma,Gesellschaft mit beschränkter Haftung, Germany). onto the tooth surfaces with White Spot Lesions using a brush, with the applicator dabbed repeatedly onto the tooth surface without contacting soft tissues. After a few minutes, a thin and clear layer is formed. A.N. will advise the patients not to brush their teeth or chew food for at least 4 hrs after treatment; during this time, soft food and liquid might be consumed.

3-Outcomes:

1. Patient satisfaction:

   H.F.& A.R will measure patient satisfaction using Visual Analogue Scale scores. The mean and standard deviation for the VAS scores of the patients recorded preoperatively, at the time of materials application, 3,6 months review for aesthetics
2. Color change assessment:

H.F.& A.R will perform visual color evaluation using the Vita Easyshade Compact (Vita Zahnfabrik, Bad Sa¨ckingen,Germany).

The shade tab may now be measured by holding the probe tip at 90° to surface at the middle 1/3 of the tab, pressing the measurement button on the Hand Piece, and waiting until the Easyshade "beeps" to indicate successful completion of the measurement H.F.& A.R will hold the probe tip 90ᴼ to the WSL on tooth surface and pressing the measurement bottom on the hand piece and waiting until the easyshade beeps to indicate successful completion of the measurement , Three images will be captured for each tooth at each time point, and the average values for L* (lightness, achromatic color coordinate), a* (green/red coordinate), b* (blue/yellow coordinate), and the resultant color difference (ϪE*) over the three measurements will be calculated H.F.& A.R will perform the visual color assessments at baseline (T0) to record the color characteristics of the WSLs immediately after treatment, (T1) to record the color characteristics of the WSL after 3 months, (T2) to record the color characteristics of the WSL after 6 months. The instrumental color measurements will be performed using the Commission International de I'Eclariage (CIE) L*a*b* color notation system (CIELAB).

ELIGIBILITY:
Inclusion Criteria:

1. No systemic disease.
2. Has completed fixed orthodontic treatment, brackets debonded.
3. Has at least two teeth with white spot lesion.
4. Has received conventional periodontal therapy after orthodontic treatment.
5. Between the ages of 12 and 25 years of age

Exclusion Criteria:

1. presence of enamel hypoplasia or dental fluorosis.
2. presence of tetracycline pigmentation.
3. periodontal pocketing of 3mm or greater.
4. taking antibiotics.
5. presence of carious cavities.
6. allergy to fluoride gel / varnish being used in study.
7. Subjects who had evidence of reduced salivary flow or significant tooth wear

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
change in patient satisfaction | before, after 3 and 6 months
  using visual analogue scale from 0-100 (0= not satisfied , 100= totally satisfied)

SECONDARY OUTCOMES:
change in color shade | before, after 3 and 6 months
  will use vita easy shade devise

IPD SHARING:
Plan to Share IPD: No